CLINICAL TRIAL: NCT03260920
Title: A Phase 2 Clinical Trial of Intranasal Oxytocin for Frontotemporal Dementia
Brief Title: Intranasal Oxytocin for Frontotemporal Dementia
Acronym: FOXY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Weston Brain Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Berry Consultants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FTDOXY17EF
Record Dates: First submitted 2017-07-19; First posted 2017-08-24 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Frontotemporal Dementia
Keywords: oxytocin; frontotemporal dementia; apathy; empathy
MeSH Terms: conditions — Frontotemporal Dementia; Lethargy | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: A Proof-of-Concept Double Blind Randomized Controlled, Cross-Over Adaptive Design Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental)
  Interventions: Drug: Syntocinon
- Medium Dose (Experimental)
  Interventions: Drug: Syntocinon
- High Dose (Experimental)
  Interventions: Drug: Syntocinon

INTERVENTIONS:
Drug: Syntocinon — Intranasal Oxytocin
  Other Names: Intranasal Oxytocin

SUMMARY:
The purpose of this study is to assess the safety, tolerability and effects on behaviour of Syntocinon given intranasally (by a spray into the nostrils) compared to placebo (an inactive saline substance that contains no medication) in participants with frontotemporal dementia/Pick's disease. This study will take place in approximately 15 centres across Canada and the United States. Approximately 112 patients in total will be enrolled in this study. In the first phase we will examine which of three different dosing schedules of oxytocin may be more effective. In the second phase of the study, patients entering the study will be randomized to the oxytocin dosing schedule that appeared most effective in the first phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable FTD (behavioural variant FTD, FTD-semantic subtype or FTD-Progressive Nonfluent Aphasia) with supportive brain imaging (centrally rated frontotemporal atrophy score of 2 or greater on brain MRI or CT) or known FTD causing genetic mutation.68
* Current symptoms of social apathy/indifference as measured by NPI apathy/indifference severity subscale score >= 2 indicating the presence of moderate to marked levels of apathy/indifference.
* Study partner who consents to study participation and who cares for/visits the patient daily for at least 3 hours/day and who can administer all trial medications.
* FTLD-CDR score 0-2.
* MMSE >10.
* Stable baseline medications related to cognition or behaviour for >=30 days such as acetylcholinesterase inhibitors, memantine, anti-depressants, antipsychotic agents, other mood stabilizers, benzodiazepines.
* Written informed consent must be obtained and documented (from the patient or, where jurisdictions allow it, from their substitute decision maker).

Exclusion Criteria:

* History of stroke, other neurologic or psychiatric disorder other than FTD that is considered to better account for behavioural symptoms.
* History of a myocardial infarction within the last two years or congestive heart failure.
* Current uncontrolled hypertension
* Current bradycardia (rate < 50 beats per minute/bpm) or tachycardia (rate > 100 bpm)
* Current hyponatremia (Na <135 mEq/L)
* Current use of topical prostaglandin medications applied to the cervix.
* Females who are pregnant or breastfeeding, or planning to conceive within the study period.
* Use of any investigational or experimental drug or device within the last 60 days prior to screening or within 5 half-lives of the experimental drug, whichever is longer.
* Participant has speech difficulties that in the opinion of the investigator would be incompatible with neuropsychology and safety assessments
* History of cancer except:

  * If considered to be cured
  * If not being actively treated with anti-cancer therapy or radiotherapy and, in the opinion of the investigator, not likely to require treatment in the ensuing 5 years
  * For prostate cancer or basal cell carcinoma, no significant progression over the previous 2 years
* Any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease. If the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
* For the CSF sub-study, current use of anticoagulant medications (warfarin, rivaroxaban, etc.).
* Plan for FTD patient to be placed into long-term care or plan for hospital admission for any kind of treatment within study period or if caregiver plans for holidays/respite care > 3 days during study period.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropsychiatric Inventory (NPI) apathy/indifference domain score | Up to 20 weeks
  Pilot data from our two prior studies of oxytocin in FTD have driven the selection of the NPI as the primary outcome measure.

SECONDARY OUTCOMES:
Change in emotional facial expression recognition performance | Up to 20 weeks
Change in the Revised Self-Monitoring Scale score | Up to 20 weeks
Change in modified Clinicians Global Impression of Change (apathy) scores | Up to 20 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - UCLA, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York
  - University of Washington, Seattle, Washington
- Canada (6):
  - University of British Columbia, Vancouver, British Columbia
  - Parkwood Institute, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Laval University, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coleman KKL, Berry S, Cummings J, Hsiung GR, Laforce R, Huey E, Ducharme S, Tartaglia MC, Mendez MF, Onyike C, Domoto-Reilly K, Masellis M, Herrmann N, Porsteinsson A, Detry MA, Stewart C, Bosse AL, McGlothlin A, Dias B, Pandey S, Mayich M, Pasternak SH, Ruiz Garcia R, Restrepo-Martinez M, Feldman H, Boxer AL, Finger EC. Intranasal oxytocin for apathy in people with frontotemporal dementia (FOXY): a multicentre, randomised, double-blind, placebo-controlled, adaptive, crossover, phase 2a/2b superiority trial. Lancet Neurol. 2025 Feb;24(2):128-139. doi: 10.1016/S1474-4422(24)00456-3. PMID 39862881
- [Derived] Finger E, Berry S, Cummings J, Coleman K, Hsiung R, Feldman HH, Boxer A. Adaptive crossover designs for assessment of symptomatic treatments targeting behaviour in neurodegenerative disease: a phase 2 clinical trial of intranasal oxytocin for frontotemporal dementia (FOXY). Alzheimers Res Ther. 2018 Sep 27;10(1):102. doi: 10.1186/s13195-018-0427-2. PMID 30261917

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT03260920/SAP_000.pdf